CLINICAL TRIAL: NCT05651672
Title: A Single-Arm Phase II Clinical Study of Pemigatinib in the Treatment of Advanced Gastrointestinal Cancer With FGFR 1-3 Alterations That Failed Standard Therapy
Brief Title: Pemigatinib in the Advanced Gastrointestinal Cancer With FGFR 1-3 Alterations
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ-0046
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Gastrointestinal Cancer
Keywords: Gastrointestinal Cancer; Pemigatinib
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — pemigatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Pemigatinib
  Interventions: Drug: Pemigatinib

INTERVENTIONS:
Drug: Pemigatinib — 13.5mg, po, 2 weeks on/1 week off, Q3W
  Other Names: Pemazyre

SUMMARY:
This study is a prospective single-arm phase II study to evaluate the efficacy and safety of Pemigatinib in the advanced gastrointestinal cancer with FGFR 1-3 alterations and failed standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Histologically or cytologically confirmed unresectable advanced, recurrent or metastatic gastrointestinal cancer
* Have at least one measurable lesion according to RECIST v1.1
* With histologically confirmed FGFR1-3 alterations, including but not limited to amplification, mutation, fusion/rearrangement
* Disease progression after prior standard therapy
* No previous use of small molecule multi-target inhibitors targeting the FGFR pathway (including but not limited to anlotinib, lenvatinib, sorafenib, apatinib)
* ECOG performance status of 0~1
* Expected survival time > 3 months
* Sufficient organ functions
* Negative pregnancy test results of childbearing age women
* Patients at risk of conception (including their partners) need to use contraception

Exclusion Criteria:

* Diagnosed with malignant tumors other than gastrointestinal cancer within 5 years before the first dose, excluding radically cured cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, and/or radically resected carcinoma in situ
* Prior receipt of selective FGFR inhibitors
* Have received any other investigational drug or participated in another interventional clinical trial within 28 days before the first dose, or have received anti-tumor drug treatment within 28 days before the first dose (including Chinese herbal medicine with anti-tumor indications)
* Have not recovered ( ≤ grade 1 or reaching the baseline, excluding asthenia and alopecia) from toxicity and/or complications caused by any intervention before the start of treatment
* Known symptomatic central nervous system metastasis and/or carcinomatous meningitis.
* Known history of allotransplantation or allogeneic hematopoietic stem cell transplantation
* Abnormal laboratory parameters listed below:

  * Serum phosphate > upper limit of normal (ULN)
  * Serum calcium exceeds the normal range, or the calcium concentration corrected for serum albumin exceeds the normal range when serum albumin exceeds the normal range
  * Potassium level < lower limit of normal (LLN)#potassium levels can be corrected by supplements at screening
* Known history of human immunodeficiency virus (HIV) infection or confirmed with positive immune test results
* Presence of severe infection in the active phase or with poor clinical control
* Pleural effusion, ascites, or pericardial effusion with obvious clinical symptoms that require drainage
* Acute or chronic active hepatitis B or C infection
* Clinically significant or uncontrolled heart diseases, including unstable angina, acute myocardial infarction within 6 months before the first dose, grade III/IV congestive heart failure (New York Heart Association), and uncontrolled arrhythmia (patients with pacemakers or with atrial fibrillation but well controlled heart rate are allowed)
* ECG changes or medical history considered clinically significant by the investigator, QTcF interval > 480 ms at screening, JTc interval can be used instead of QTc interval (in such cases, JTc must be ≤ 340 ms) for patients with intraventricular conduction block (QRS interval > 120 ms)
* Uncontrolled hypertension (systolic pressure > 160 mmHg or diastolic pressure > 100 mmHg) after the optimal medical treatment, or a history of hypertensive crisis or hypertensive encephalopathy
* Hepatic encephalopathy, hepatorenal syndrome, or liver cirrhosis with Child-Pugh grade B or C
* Have received a major surgery (craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to the first dose, or will receive a major surgery during the study treatment period
* Not fully recovered from toxicity and/or complications of a major surgery before the study treatment
* Pregnant or lactating women, or patients expected to conceive or give birth during the study period from the screening to the completion of the safety follow-up visit (90 days after the last dose for male subjects)
* Have received radiotherapy within 4 weeks before the first dose.
* History of disorders of calcium and phosphorus metabolism or systemic electrolyte metabolism imbalance with ectopic calcification of soft tissues (excluding calcification of soft tissues such as skin, kidneys, tendon, or blood vessels without systemic electrolyte metabolism imbalance caused by injury, disease, and old age)
* Clinically significant corneal or retinal diseases confirmed by ophthalmological examination
* Prior receipt of any potent CYP3A4 inhibitor or inducer within 14 days or 5 half lives (whichever is shorter) before the first dose. Ketoconazole is allowed for external use
* Known allergic reactions to pemigatinib or excipients of pemigatinib
* Unable or unwilling to swallow pemigatinib or are suffering from significant digestive system diseases that may interfere with absorption, metabolism, or excretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | up to 2 years
  Defined as proportion of patients who have a best response of complete response (CR) + partial response (PR) according to the RECIST 1.1 criteria

SECONDARY OUTCOMES:
Progress Free Survival (PFS) | Up to 4 years
  Defined as the time from enrollment to disease progression or death (whichever occurs first)
Overall Survival (OS) | Up to 4 years
  Defined as the time from enrollment to the death
Duration of Response (DOR) | up to 4 years
  Defined as the time from the date of CR or PR to PD
Disease Control Rate (DCR) | Up to 2 years
  Defined as proportion of patients who have a best response of complete response (CR) + partial response (PR) + stable disease (SD) according to the RECIST1.1 criteria
Adverse Events (AEs) | Up to 2 years
  Defined as the proportion of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), serious adverse event (SAE), assessed by NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China